CLINICAL TRIAL: NCT05190666
Title: Physical Activity and Weight Loss to Improve Function and Pain After Total Knee Replacement
Brief Title: Healthy Living After Knee Replacement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Christine A Pellegrini, PhD, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00109459; R01AG070004 (NIH)
Record Dates: First submitted 2021-12-28; First posted 2022-01-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Arthroplasty; Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PACE Weight Loss Program (Experimental): Participants randomized to this arm will receive personalized diet, activity, and weight loss goals as well as tools to self-monitor behaviors and weight. To facilitate changes, participants will receive coaching calls weekly during months 1-4, biweekly during months 5-6, and monthly during months 7-12.
  Interventions: Behavioral: PACE Weight Loss program
- Chronic Disease Self-Management Program (Sham Comparator): Participants randomized to this arm will receive a chronic disease self-management program including a self-management book. Participants will receive regular calls weekly during months 1-4, biweekly during months 5-6, and monthly during months 7-12.
  Interventions: Behavioral: Chronic Disease Self-Management

INTERVENTIONS:
Behavioral: PACE Weight Loss program — 12 month phone-based behavioral weight loss program
  Arms: PACE Weight Loss Program
Behavioral: Chronic Disease Self-Management — 12 month phone-based chronic disease self-management program
  Arms: Chronic Disease Self-Management Program

SUMMARY:
The purpose of this study is to examine if a weight loss program designed for adults after knee replacement improves weight loss, physical activity, pain, and function, as well as if the program is cost effective, as compared to a chronic disease self-management program.

DETAILED DESCRIPTION:
Participants will be randomized to either a weight loss program or chronic disease self-management program. Both programs will be phone-based and include phone calls with a health coach weekly during months 1-4, biweekly during months 5-6, and monthly during months 7-12. Monthly calls with occur between months 13-18. Assessments examining outcomes will be completed at baseline, 6, 12, and 18 months.

ELIGIBILITY:
Inclusion Criteria:

Participants must:

* have a body mass index between 25-45 kg/m2
* have had a knee replacement (including primary, staged or independent bilateral, or revision) <6 months prior to baseline assessment
* have a computer, tablet, or smartphone with active internet access to self-monitor online and/or have a device or computer compatible with Fitbit
* completion of baseline assessment measures (height, weight, function tests, surveys, ≥4 days valid of activity monitoring, and 1 day of dietary recall)
* be English-speaking and able to read consent and study materials written in English
* be willing to attend 4 in-person assessments.

Exclusion Criteria:

* have any contraindications to diet or weight loss
* undergo simultaneous bilateral knee replacement or have a scheduled or anticipated knee replacement for the contralateral knee within the next 18 months
* have a mobility limiting comorbidity unrelated to knee replacement (e.g. spinal stenosis, fibromyalgia, peripheral vascular disease, stroke)
* are taking anti-obesity medications
* are enrolled in a formal weight loss program
* had or are planning to have bariatric/gastric/lap band surgery
* are planning to relocate out of the Columbia or Greenville, SC areas in the next 18 months.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in body weight at 6 months | 6 months
  kg

SECONDARY OUTCOMES:
Change in WOMAC pain subscale at 6 months | 6 months
  WOMAC Pain Subscale - Scores range from 0 (no pain) to 20 (maximal pain)
Change in WOMAC pain subscale at 12 months | 12 months
  WOMAC Pain Subscale - Scores range from 0 (no pain) to 20 (maximal pain)
Change in WOMAC pain subscale at 18 months | 18 months
  WOMAC Pain Subscale - Scores range from 0 (no pain) to 20 (maximal pain)
Change in Six Minute Walk Duration at 6 months | 6 months
  Physical function assessed with the six minute walk test (feet)
Change in Six Minute Walk Duration at 12 months | 12 months
  Physical function assessed with the six minute walk test (feet)
Change in Six Minute Walk Duration at 18 months | 18 months
  Physical function assessed with the six minute walk test (feet)
Change in Timed Up & Go at 6 months | 6 months
  Physical function assessed with the Timed Up & Go Test (seconds)
Change in Timed Up & Go at 12 months | 12 months
  Physical function assessed with the Timed Up & Go Test (seconds)
Change in Timed Up & Go at 18 months | 18 months
  Physical function assessed with the Timed Up & Go Test (seconds)
Change in Chair Stands at 6 months | 6 months
  Physical function assessed with the Chair stand test (# of chair stands)
Change in Chair Stands at 12 months | 12 months
  Physical function assessed with the Chair stand test (# of chair stands)
Change in Chair Stands at 18 months | 18 months
  Physical function assessed with the Chair stand test (# of chair stands)
Change in Moderate to vigorous intensity physical activity at 6 months | 6 months
  Objectively measured by Actigraph accelerometer (>=2020 counts/min)
Change in Moderate to vigorous intensity physical activity at 12 months | 12 months
  Objectively measured by Actigraph accelerometer (>=2020 counts/min)
Change in Moderate to vigorous intensity physical activity at 18 months | 18 months
  Objectively measured by Actigraph accelerometer (>=2020 counts/min)
Change in body weight at 12 months | 12 months
  kg
Change in body weight at 18 months | 18 months
  kg

CONTACTS AND LOCATIONS:
Overall Officials: Christine Pellegrini, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
We will also make de-identified study data available 12 months after the primary manuscript is published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months after primary manuscript is published
Access Criteria: Open